CLINICAL TRIAL: NCT05409755
Title: Efficacy of Fractional Needling Radiofrequency in Female Pattern Hair Loss, a Randomized Controlled Trial.
Brief Title: Radiofrequency in Female Pattern Hair Loss
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hagar El Sayed, Dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Female pattern hair loss
Record Dates: First submitted 2022-05-20; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Female Pattern Baldness
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fractional microneedling radiofrequency (Active Comparator): Device
  Interventions: Other: Vivacy
- Fractional microneedling radiofrequency followed by minoxidil application (Active Comparator): Device and drug
  Interventions: Other: Vivacy
- Minoxidil (Active Comparator): Topical drug
  Interventions: Other: Vivacy

INTERVENTIONS:
Other: Vivacy — Vivacy and minoxidil

SUMMARY:
Pattern hair loss, also called androgenetic alopecia (AGA) is considered the most common cause of hair loss in both males and females affecting approximately 85% of males and 50% of females over 50 years of age.

DETAILED DESCRIPTION:
RF (Radiofrequency) based devices have also been shown to be successful in promoting hair growth, thought to occur through the induction of growth factors in the papillary dermis. Studying the effect of fractional needling radiofrequency in the treatment of female pattern hair loss will pave the way for more treatment options for this common disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with female pattern hair loss

Exclusion Criteria:

* - Pregnancy and lactation.
* Bleeding tendency.
* Cases who received treatment (systemic or topical) in the last 3 months before treatment.
* Scarring alopecia.
* Other associated causes of alopecia

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-25 (Estimated); Primary Completion 2022-09-15 (Estimated); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
Clinical examination by Sinclair scale | 3 months
  Clinical